CLINICAL TRIAL: NCT01645436
Title: Physical Activity in Pediatric Cancer Patients With Solid Tumor Trial
Brief Title: Physical Activity in Pediatric Cancer (PAPEC)
Acronym: PAPEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Alejandro Lucia, MD PhD, PROFESSOR IN EXERCISE PHYSIOLOGY, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LUCIA
Record Dates: First submitted 2012-07-15; First posted 2012-07-20 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Pediatric Cancer
Keywords: randomized controlled trial; in-hospital exercise; children; cancer
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (exercise) (Experimental): combined inpatient physical training (aerobic + strength) over neoadjuvant chemotherapy. The intervention will include three weekly exercise sessions of 60-90 minutes, and will be held in child's room or in a pediatric gym specifically enabled on the aforementioned hospital, depending on the children's health status.
  Interventions: Other: exercise training
- control (usual care) (No Intervention): Usual hospital care with no exercise

INTERVENTIONS:
Other: exercise training — The intervention group will participate in combined inpatient physical training (aerobic + strength) over neoadjuvant chemotherapy. The intervention will include three weekly exercise sessions of 60-90 minutes, and will be held in child's room or in a pediatric gym specifically enabled on the aforementioned hospital, depending on the children's health status.
  Other Names: physical activity
  Arms: treatment (exercise)

SUMMARY:
The aim of this randomized controlled trial on Physical Activity and Pediatric Cancer (PAPEC) is to assess the impact of an exercise program intervention in pediatric cancer patients undergoing chemotherapy for solid tumors. The investigators hypothesized the intervention will have a beneficial effect on the study outcomes.

DETAILED DESCRIPTION:
Sixty patients, of both sexes, children will be recruited for this trial with an age range between 4 to 16 years old, undergoing treatment for primary tumors (excluding central nervous system tumors). Each participant will be assigned randomly (with blocking on sex) to either intervention or control (usual care) group.

The intervention group will participate in combined inpatient physical training (aerobic + strength) over neoadjuvant chemotherapy. The intervention will include three weekly exercise sessions of 60-90 minutes, and will be held in child's room or in a pediatric gym specifically enabled on the aforementioned hospital, depending on the children's health status.

Primary outcomes [cardio-respiratory capacity (peak oxygen uptake), muscle strength (6RM leg and bench press, and lateral row), functional capacity ('Timed Up and Down Stairs test', and '3 m and 10m Time Up and Go tests'), physical activity levels (determined by accelerometry) and quality of life "Child Report Form of the Child's Health and Illness Profile-Child Edition", Adolescent Edition and Parents Report Form )] and secondary outcomes [immune function (immune cell subpopulations, natural killer cells' cytotoxicity), inflammatory profile (blood levels of 47 cytokines) and leukocyte telomere length] will be measured in both groups in the following time points:

(i) before the exercise intervention (immediately after diagnosis and before the start of treatment); (ii) after the exercise intervention (upon termination of neoadjuvant chemotherapy); and iii) after a detraining period (2 months after the intervention).

ELIGIBILITY:
Inclusion Criteria:

* age range between 4 to 16 years old, undergoing treatment for primary tumors (excluding central nervous system tumors) treated in the Hospital Infantul Niño jesús and residents in Madrid community. -

Exclusion Criteria:

* age<4 years or >16 years, other tumours

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Muscle strength (kg) measured in 5-repetition maximum (5RM) leg and bench press and lateral row exercise tests | up to 3 years

SECONDARY OUTCOMES:
inflammatory profile | up to 3 years
  blood levels of 47 cytokines (including, among others, interferon (IFN) α2, IFNγ, interleukin (IL)1α, IL1ß, IL1ra, IL2, IL2RA, IL3, IL4, IL6, IL7, IL8, IL9, IL10, IL12, IL13, IL15, IL16, IL17, tumor necrosis factor(TNF)-related apoptosis-inducing ligand, and TNFα.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Lucia, MD PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Soares-Miranda L, Fiuza-Luces C, Lassaletta A, Santana-Sosa E, Padilla JR, Fernandez-Casanova L, Lorenzo-Gonzalez R, Lopez-Mojares LM, Perez M, Perez-Martinez A, Lucia A. Physical Activity in Pediatric Cancer patients with solid tumors (PAPEC): trial rationale and design. Contemp Clin Trials. 2013 Sep;36(1):106-15. doi: 10.1016/j.cct.2013.05.012. Epub 2013 Jun 5. PMID 23747802